CLINICAL TRIAL: NCT03647540
Title: The Application of Fluorescence Laparoscopy in the Treatment of Adenocarcinoma of the Esophagogastric Junction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dong Yang (Other)
Responsible Party: Sponsor-Investigator, Dong Yang, Doctor, Jilin University
Organization: Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 130020
Record Dates: First submitted 2018-08-23; First posted 2018-08-27 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Fluorescence Laparoscopy; Adenocarcinoma of the Esophagogastric Junction
Keywords: fluorescence laparoscopy; adenocarcinoma of the esophagogastric junction (AEG)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group F (Experimental): Group F received endoscopic submucosal injection of indocyanine green (ICG) 2 hours before operation, followed by fluorescent laparoscopic radical gastrectomy. All specimens were grouped for lymph node collection, and the postoperative management was unified according to enhanced recovery after surgery (ERAS). All basic clinical and pathological data were statistically analyzed
  Interventions: Procedure: fluorescent laparoscopic radical gastrectomy
- Group L (Active Comparator): Group L received traditional laparoscopic radical gastrectomy. All specimens were grouped for lymph node collection, and the postoperative management was unified according to enhanced recovery after surgery (ERAS). All basic clinical and pathological data were statistically analyzed
  Interventions: Procedure: traditional laparoscopic radical gastrectomy

INTERVENTIONS:
Procedure: fluorescent laparoscopic radical gastrectomy — The gastrectomy for group F would be underwent by the fluorescence laparoscopy. All surgical procedures will be performed by the surgery team ,which is leaded by professor Wang Quan.
  Arms: Group F
Procedure: traditional laparoscopic radical gastrectomy — The gastrectomy for group L would be underwent by the laparoscopy.All surgical procedures will be performed by the surgery team ,which is leaded by professor Wang Quan.
  Arms: Group L

SUMMARY:
The fluorescent laparoscopic technique would be applied to the radical resection of gastric cancer at the junction of esophagus and stomach, and compared with the traditional laparoscopic radical resection of gastric cancer to find a better surgical method for patients

ELIGIBILITY:
Inclusion Criteria:

- 1. All cases should be diagnosed as adenocarcinoma of the esophagogastric junctionncer by histology. The tumor is within 1 cm above or 2 cm below the anatomic cardia. The clinical stage is T1-3, Nx, M0 for gastric cancer which can undergo the laparoscopic surgery.

2. Eastern Cooperative Oncology Group (ECOG) scale 0-2 3. Heart, lung, liver, and kidney function can tolerate operation 4. Patients and their families are able to understand and be willing to participate in this clinical study and to sign informed consent.

Exclusion Criteria:

1. history of stomach malignant disease 2. recent diagnosis of other malignant tumors (except for papillary carcinoma of the thyroid gland and basal cell carcinoma of the skin) 3. patients with obstruction, perforation, bleeding requiring emergency surgery 4. a history of abdominal surgery (which makes it difficult to perform laparoscopic procedures), severe systemic disease such as diabetes, severe chronic lung disease, cirrhosis, other malignant diseases 5. combined stomach multiple carcinomas 6. with a history of serious mental illness 7. pregnant or lactating women 8. The researchers believe that the patients are unsuitable to participate in the researchers with other cases.

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2018-08-30 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
the number of the dissected lymph nodes | in the perioperative period
  It includes the total number of the dissected lymph nodes and every group of lymph nodes

SECONDARY OUTCOMES:
3-year disease-free survival | three years after operation]
the incidence of complications | one month after surgery
the operation time | in the perioperative period
  The descriptive name of unit would be minute (min).
the blood loss during the operation | in the perioperative period
  The descriptive name of unit would be millilitre (ml).
Postoperative recovery of intestinal peristalsis | in the perioperative period
  The descriptive name of unit would be hour (h).
cases converted to open surgery | in the perioperative period
The mean postoperative hospital stay | in the perioperative period
  The descriptive name of unit would be day (d).

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hospital of Jilin University, Ch’ang-ch’un, Jilin, China

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.